CLINICAL TRIAL: NCT00688831
Title: A Single-centre, Single-blind, Randomised, Placebo-controlled, Single-dose Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics After Ascending Intravenous Doses of AZD1305 in Helahty Male Volunteers
Brief Title: Single Ascending Dose Study (SAD) iv Formulation
Acronym: 2006-006253-27
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrythmias & Lipids, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3190C00002
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: AZD1305; SAD; safety; pharmcokinetics; Safety and tolerability
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD1305 solution for iv infusion
  Interventions: Drug: AZD1305
- B (Placebo Comparator): NaCl solution for iv infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — Solution for iv infusion , single dose
  Arms: A
Drug: Placebo — NaCl solution for iv infusion, single dose
  Arms: B

SUMMARY:
The purpose is to study the safety of AZD1305, how AZD1305 is tolerated and how the medication is metabolised by the body (how it is taken up into the body, distributed around the body and disappears from the body

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BIM 19-30 kg/m2

Exclusion Criteria:

* Potassium outside normal reference values
* ECG findings outside normal range

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Adverse events, ECG variables, vital signs, physical examination, laboratory variables, body temperature and weight | During the study

SECONDARY OUTCOMES:
Pharmacokinetic variables | During all dosing visits

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Marianne Hartford, MD, PhD, Principal Investigator — AstraZeneca, Clinical Pharmacology Unit, Sahlgrenska University Hospital, Göeborg, Sweden
Locations (1):
- Research Site, Uppsala, Sweden